CLINICAL TRIAL: NCT00704314
Title: Effects of High Dose Simvastatin Therapy on Glucose Metabolism and Ectopic Lipid Deposition in Non-Obese Type 2 Diabetic Patients
Brief Title: Does Simvastatin Affect Insulin Sensitivity in Dyslipidemic Type 2 Diabetic Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Austrian Science Fund (FWF) (Other); European Foundation for the Study of Diabetes (Other); EU grant (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Prof. Dr. Werner Waldhäusl, Prof. Dr. Michael Roden, Hanusch Hospital, 1. Medical Department, Vienna Austria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EK: 258/2002
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Hypercholesterolemia; Diabetes; Cardiovascular Disease
Keywords: Insulin resistance; Statins; Muscle and liver triglycerides
MeSH Terms: conditions — Hypercholesterolemia; Diabetes Mellitus; Cardiovascular Diseases; Insulin Resistance | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Simvastatin therapy, 80 mg/d for 8 weeks
  Interventions: Drug: Simvastatin
- 2 (Placebo Comparator): Placebo, one pill daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — 80 mg Simvastatin daily for 8 weeks
  Other Names: Zocord
  Arms: 1
Drug: Placebo — The placebo was identical in appearance and was provided by the same manufacturer
  Arms: 2

SUMMARY:
We aimed to address the issue whether statins affect insulin resistance. To this end, we combined the available state-of-the art technology for detailed assessment of both whole-body and tissue specific insulin sensitivity in vivo in humans (euglycemic-hyperinsulinemic clamp, stable isotope [6,6-2H2]glucose dilution technique, proton nuclear magnetic resonance spectroscopy - 1H MRS - of liver and skeletal muscle). Outcome measures were determined before and after 8 weeks therapy with 80 mg Simvastatin in hypercholesterolemic patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with known duration of disease: 3-10 years
* Age: 35-75 years
* BMI<32 kg/m2
* Hypercholesterolemia: fasting serum low density lipoprotein (LDL)
* Cholesterol concentration < 4.16 mmol/L (<160 mg/dl)
* Normotriglyceridemia: fasting plasma triglyceride concentration < 2.75 mmol/L (250 mg/dl)
* Creatinine levels < 1.8 mg /dl
* Liver transaminases < 20% over the upper limit with no active liver disease and CK < 50% above the upper limit
* Blood pressure less than 160/100 mmHg were accepted as eligible for enrollment

Exclusion Criteria:

* Hypertension, cardiovascular disease or metabolic diseases other than T2DM as determined by medical history, physical examination and routine laboratory tests
* Alcohol consumption (more than 10 drinks/week)
* Poor glycemic control (HbA1c<9%)
* Patients requiring insulin, patients with type 1 diabetes
* Patients taking any medicine known to interfere with metabolism of statins or with insulin sensitivity as summarized in an exclusionary drug table
* Patients receiving any hypolipidemic medication or diet during the last 2 months before enrollment

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-10; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | 8 weeks

SECONDARY OUTCOMES:
ectopic lipid deposition in liver and muscle | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Werner Waldhäusl, Prof, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Szendroedi J, Anderwald C, Krssak M, Bayerle-Eder M, Esterbauer H, Pfeiler G, Brehm A, Nowotny P, Hofer A, Waldhausl W, Roden M. Effects of high-dose simvastatin therapy on glucose metabolism and ectopic lipid deposition in nonobese type 2 diabetic patients. Diabetes Care. 2009 Feb;32(2):209-14. doi: 10.2337/dc08-1123. Epub 2008 Oct 28. PMID 18957532